CLINICAL TRIAL: NCT07360587
Title: Thyroid Artery Embolization for the Treatment of Compressive Goiters: a Prospective Cohort Study.
Brief Title: Thyroid Artery Embolization for the Treatment of Compressive Goiters.
Acronym: TAE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Laurent Fradet, MD, FRCSC, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-5830
Record Dates: First submitted 2025-12-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Nodules
Keywords: Goiter; Thyroid Artery Embolization; thyroid nodule
MeSH Terms: conditions — Thyroid Nodule; Goiter

STUDY DESIGN:
Intervention Model Description: This study is a prospective interventional cohort study. The prospective cohort setting allows us to evaluate the direct effect of TAE on a series of patients on a longer period and to strengthen the retrospective data previously documented in other studies. There is no comparative group in our study as it aims to prove that TAE is effective and safe in a "nonsurgical" population, a population in which other alternatives lack or are refused by the patient.
Masking Description: No needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thyroid Artery Embolization (Experimental): Patients with diagnosis of Goiter with compressive symptoms in which other alternatives lack or are refused by the patient himself.
  Interventions: Procedure: Thyroid Artery Embolization

INTERVENTIONS:
Procedure: Thyroid Artery Embolization — Interruption of blood flow that supplies thyroid nodule using embolization technique.

SUMMARY:
Very few studies have investigated TAE as a treatment for goiter with compressive symptoms. What is the efficacy and safety of TAE for the treatment of compressive goiters in a population ineligible for or refusing standard therapy? This is a prospective interventional cohort study that will allow us to standardize imaging by improving quality data collection and fellow-up to assess the efficacy of TAE for compressive symptoms of nodular goiters. Not only to corroborate current emerging results but clearly define the expected results for this technique.

DETAILED DESCRIPTION:
This study is a prospective interventional cohort study.

The prospective cohort setting allows us to evaluate the direct effect of TAE on a series of patients on a longer period and to strengthen the retrospective data previously documented in other studies.

Included patients will have compressive symptoms or significant tracheal or oesophageal compression at risk of causing symptoms attributed to a goiter.

They have to be Ineligible for surgery/ablative treatments or preference for TAE over other treatments.

There is no comparative group in our study as it aims to prove that TAE is effective and safe in a "nonsurgical" population, a population in which other alternatives lack or are refused by the patient.

Our sampling method will be a non-probabilistic convenience sampling. Patients will be recruited in an outpatient setting by the patient's treating endocrinologist or otolaryngologist.

ELIGIBILITY:
Inclusion Criteria:

* Patient with compressive symptoms or significant tracheal or oesophageal compression at risk of causing symptoms attributed to a goiter AND
* Ineligible for surgery/ablative treatments or preference for TAE over other treatments AND
* TiRADS category 1, 2, 3 or 4 AND
* Bethesda categories I or III on 2 different biopsies OR Bethesda II on one biopsy AND
* Patient at least 18 years old.

Exclusion Criteria:

* Comorbidities precluding endovascular procedure OR
* TiRADS category 5 OR
* Bethesda categories IV, V, VI on biopsy OR
* Refusal of the patient to participate OR
* Uncontrolled severe hyperthyroidism OR
* Minor patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Thyroid nodule volume | Follow-ups at 1 week, and 3 months, 6 months and 12 months post-op.
  TAE effectiveness to reduce overall thyroid and nodular volumes in benign compressive goiters assessing changes in Nodule(s) volume(s) and Thyroid lobe volume.

SECONDARY OUTCOMES:
Change in symptoms after TAE. | Follow-ups at 3 months, 6 months and 12 months post-op.
  Assess the impact of TAE on the symptoms related to the goiter as reported by the patient. Using ThyPRO score.
  ThyPRO is designed to evaluate physical, psychological, and social impairments caused by benign thyroid diseases by evaluating :
  * Symptom severity
  * Functional limitations
  * Emotional and social impacts
  * This disease-specific focus supports patient-centered care, clinical decision-making, and outcomes research.
  * Target Population ThyPRO is validated for adults aged 18 and older with benign thyroid diseases.
  The ThyPRO consists of 85 items, grouped into:
  13 multi-item domains: Goiter symptoms (11 items) Hyperthyroid symptoms (8) Hypothyroid symptoms (4) Eye symptoms (8) Tiredness (7) Cognitive impairment (6) Anxiety (6), Depressivity (7) Emotional susceptibility (9) Impaired social life (4), daily life (6), and sex life (2) Cosmetic complaints (6)
  1 global QoL item Each question is rated on a 5-point Likert scale (0 = Not at all to 4 = Completely
Safety level of TAE in compressive goiter: Adverse Events report | Day of embolisation; Follow-ups at 1 week, and 3 months, 6 months and 12 months post-op.
  Evaluate the safety of TAE for the treatment of benign compressive goiter using the Adverse Events report.
Safety level of TAE in compressive goiter: thyroid function tests | At baseline visit, approximately 48 hours after the intervention, and 6 weeks, 3 months, 6 months and 12 months after the intervention. More tests can be done according to the treating physician.
  Monitoring of the effect of the intervention with thyroid function tests.
Safety level of TAE in compressive goiter: parathyroid function tests | At baseline visit, approximately 48 hours after the intervention, and 6 weeks, 3 months, 6 months and 12 months after the intervention. More tests can be done according to the treating physician.
  Describe the effect of the procedure on parathyroid function with PTH and calcium blood levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
IPD information will only be shared after a formal request sent to the principal investigator's email address if the latter considers that the request is legally scientifically justified.

REFERENCES:
- [Background] Ramos HE, Braga-Basaria M, Haquin C, Mesa CO, Noronha Ld, Sandrini R, Carvalho Gde A, Graf H. Preoperative embolization of thyroid arteries in a patient with large multinodular goiter and papillary carcinoma. Thyroid. 2004 Nov;14(11):967-70. doi: 10.1089/thy.2004.14.967. PMID 15671777
- [Background] Bonnici M, Nevin C, Boo S. Thyroid ima artery embolization for the treatment of Graves' disease and thyroid storm. Radiol Case Rep. 2023 May 28;18(8):2641-2644. doi: 10.1016/j.radcr.2023.04.044. eCollection 2023 Aug. PMID 37273723
- [Background] Xiao H, Zhuang W, Wang S, Yu B, Chen G, Zhou M, Wong NC. Arterial embolization: a novel approach to thyroid ablative therapy for Graves' disease. J Clin Endocrinol Metab. 2002 Aug;87(8):3583-9. doi: 10.1210/jcem.87.8.8723. PMID 12161479
- [Background] Galkin EV, Grakov BS, Protopopov AV. [First clinical experience of radio-endovascular functional thyroidectomy in the treatment of diffuse toxic goiter]. Vestn Rentgenol Radiol. 1994 May-Jun;(3):29-35. Russian. PMID 7985368
- [Background] McDermott MT. Hyperthyroidism. Ann Intern Med. 2020 Apr 7;172(7):ITC49-ITC64. doi: 10.7326/AITC202004070. PMID 32252086
- [Background] Lim HK, Lee JH, Ha EJ, Sung JY, Kim JK, Baek JH. Radiofrequency ablation of benign non-functioning thyroid nodules: 4-year follow-up results for 111 patients. Eur Radiol. 2013 Apr;23(4):1044-9. doi: 10.1007/s00330-012-2671-3. Epub 2012 Oct 25. PMID 23096937
- [Background] Guan SH, Wang H, Teng DK. Comparison of ultrasound-guided thermal ablation and conventional thyroidectomy for benign thyroid nodules: a systematic review and meta-analysis. Int J Hyperthermia. 2020;37(1):442-449. doi: 10.1080/02656736.2020.1758802. PMID 32369708
- [Background] Papini E, Gugliemi R, Pacella CM. Laser, radiofrequency, and ethanol ablation for the management of thyroid nodules. Curr Opin Endocrinol Diabetes Obes. 2016 Oct;23(5):400-6. doi: 10.1097/MED.0000000000000282. PMID 27504993
- [Background] Haugen BR, Alexander EK, Bible KC, Doherty GM, Mandel SJ, Nikiforov YE, Pacini F, Randolph GW, Sawka AM, Schlumberger M, Schuff KG, Sherman SI, Sosa JA, Steward DL, Tuttle RM, Wartofsky L. 2015 American Thyroid Association Management Guidelines for Adult Patients with Thyroid Nodules and Differentiated Thyroid Cancer: The American Thyroid Association Guidelines Task Force on Thyroid Nodules and Differentiated Thyroid Cancer. Thyroid. 2016 Jan;26(1):1-133. doi: 10.1089/thy.2015.0020. PMID 26462967
- [Background] Khairy GA. Solitary thyroid nodule: the risk of cancer and the extent of surgical therapy. East Afr Med J. 2004 Sep;81(9):459-62. doi: 10.4314/eamj.v81i9.9221. PMID 15626055
- [Background] Guth S, Theune U, Aberle J, Galach A, Bamberger CM. Very high prevalence of thyroid nodules detected by high frequency (13 MHz) ultrasound examination. Eur J Clin Invest. 2009 Aug;39(8):699-706. doi: 10.1111/j.1365-2362.2009.02162.x. PMID 19601965